CLINICAL TRIAL: NCT04240223
Title: A Phase 1, Single Dose Escalation Study to Investigate the Use of Delayed Release Tablets for Colonic Delivery of Brilacidin in Healthy Volunteers
Brief Title: A Study to Investigate the Use of Delayed Release Tablets for Colonic Delivery of Brilacidin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovation Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: BC250; 2019-003367-22 (EudraCT Number)
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — brilacidin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 50 mg Brilacidin tablet (Experimental)
  Interventions: Drug: Brilacidin; Radiation: 4Mq 99mTc-DTPA
- 100 mg Brilacidin tablet (Experimental)
  Interventions: Drug: Brilacidin; Radiation: 4Mq 99mTc-DTPA
- 200 mg Brilacidin (2 x 100 mg Brilacidin tablets) (Experimental)
  Interventions: Drug: Brilacidin; Radiation: 4Mq 99mTc-DTPA
- Placebo tablet (replica of shape/size of 50 mg tablet) (Placebo Comparator)
  Interventions: Drug: Placebo; Radiation: 4Mq 99mTc-DTPA
- Placebo tablet (replica of shape/size of 100 mg tablet) (Placebo Comparator)
  Interventions: Drug: Placebo; Radiation: 4Mq 99mTc-DTPA
- Placebo (2 x replica of shape/size of 100 mg tablets) (Placebo Comparator)
  Interventions: Drug: Placebo; Radiation: 4Mq 99mTc-DTPA

INTERVENTIONS:
Drug: Brilacidin — Brilacidin
  Arms: 100 mg Brilacidin tablet; 200 mg Brilacidin (2 x 100 mg Brilacidin tablets); 50 mg Brilacidin tablet
Drug: Placebo — Placebo
  Arms: Placebo (2 x replica of shape/size of 100 mg tablets); Placebo tablet (replica of shape/size of 100 mg tablet); Placebo tablet (replica of shape/size of 50 mg tablet)
Radiation: 4Mq 99mTc-DTPA — 4Mq technetium-99m (99mTc), complexed with diethylenetriaminepentaacetic acid (DTPA) which prevents absorption of the radioisotope from the gastrointestinal tract

SUMMARY:
This is a single-centre, blinded, randomized, placebo controlled, dose escalation study. Up to 9 healthy male volunteers will participate in the study. This study is designed to investigate the use of delayed release tablets for colonic delivery of Brilacidin.

DETAILED DESCRIPTION:
Brilacidin is a fully synthetic, non-peptidic, host defense protein mimetic, and has been shown to demonstrate anti-inflammatory and antibacterial activities.

Two prototype tablets have been developed to contain 50 mg or 100 mg of Brilacidin. Matching placebo tablets have also been developed. In this Phase 1 study, the delayed release prototype tablets will be tested to confirm efficient and specific target release of Brilacidin in the colon and to assess the safety, tolerability and the pharmacokinetics of Brilacidin administered directly to the colon.

Three subjects will be enrolled into each cohort of the study. Each subject will receive one treatment at one Assessment Visit. In each cohort, two subjects will receive a Brilacidin containing dose, and one subject will receive placebo.

Cohort 1: 50 mg Brilacidin or Placebo; Cohort 2: 100 mg Brilacidin or Placebo; Cohort 3: 200 mg Brilacidin (as 2 x 100 mg Brilacidin tablets) or 2 x Placebo.

Each treatment (drug and placebo) will be radiolabelled with technetium-99m (99mTc). The radiopharmaceutical, 99mTc-DTPA, does not enter the systemic circulation and is routinely used for investigations of this type. In Cohort 1 and 2 each tablet, including placebo, will be radiolabelled to contain approximately 4 MBq 99mTc-DTPA at time of dosing. In Cohort 3 each individual tablet, active or placebo, will be radiolabelled with 2 MBq 99mTc-DTPA to give a total dose of 4 MBq per treatment.

Each tablet will be taken orally with 200 mL room temperature water with subjects in the fasted state. The gastrointestinal transit and release behavior of the tablets will be studied using gamma scintigraphy. Blood samples will be taken at pre-defined times to allow pharmacokinetic (PK) evaluation of drug absorption with respect to time and location of tablet release.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers.
2. Aged between 18 and 65 years inclusive.
3. BMI between 18 and 30 kg/m², inclusive. Body weight ≥50 kg.
4. Understands and is willing, able and likely to comply with all study procedures and restrictions.
5. Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent (signed and dated) obtained before any trial-related activities.
6. Confirmed to be in general good health.

Exclusion Criteria:

1. Medical History

   1. Current or recurrent disease that, in the opinion of the PMI or medically qualified designee/physician responsible, could affect the study conduct or laboratory assessments (e.g. hepatic disorders, renal insufficiency, congestive heart failure).
   2. Current or relevant previous history of serious, severe or unstable physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that presents undue risk from the study medication or procedures.
   3. A history of current or relevant previous non self-limiting gastrointestinal disorders.
   4. Currently suffering from disease known to impact gastric emptying, e.g. migraine, Type 1 or Type 2 diabetes mellitus.
   5. Has untreated hypertension or has hypertension under treatment.
   6. Has a diagnosis of an immunosuppressive illness or a condition requiring chronic immunosuppression.
   7. As a result of physical examination or screening investigations, and available prior to dosing evaluations, the PMI or medically qualified designee/ physician responsible considers the volunteer unfit for the study.
2. Medications

   1. Subject is scheduled to take prescribed medication within 14 days prior to the assessment visit.
   2. Subject is scheduled to take over-the-counter (OTC) medication, including vitamins and natural or herbal remedies, within 48 hours prior to the assessment visit.
3. Alcohol/Substance Abuse

   1. Recent history (within the last year) of alcohol or other substance abuse.
   2. Subject has an average weekly alcohol intake of greater than 21 units.
   3. Subject has positive urine drugs of abuse test at screening or prior to dosing evaluation.
   4. Subject has a positive breath alcohol test at screening or prior to dosing evaluation.
4. Smoking

   1. Subject has recently discontinued smoking (less than 3 months).
   2. Subject is currently a smoker or user of nicotine-containing products.
   3. Subject has a positive urine cotinine test at screening or prior to dosing evaluation.
5. Allergy/Intolerance

   1. Subject has a history of allergy to any component of the dosage form or any other allergy, which, in the opinion of the PMI or medically qualified designee/ physician responsible, contraindicates their participation.
   2. Has known allergies or intolerance to Brilacidin.
   3. Has an allergy to any of the contents of the standardised meals.
   4. Vegetarian or vegan.
   5. Suspected or diagnosed lactose intolerance.
6. Clinical Studies

   1. Participation in another clinical study (inclusive of final post-study examination) or receipt of an investigational drug within the 12 weeks before first screening visit.
   2. Previous participation in this study.
   3. Subject whose participation in this study will result in a participation in more than four studies over a twelve month period.
7. Personnel; An employee of the Sponsor, client or study site or members of their immediate family.
8. Radiation Exposure; Subject has a total dosimetry value which, in the opinion of the PMI or medically qualified designee/ physician responsible, contraindicates their participation.
9. Blood

   1. Blood donation or significant blood loss within 3 months of screening.
   2. Difficulty accessing forearm veins for cannulation or blood sampling.
10. Family Planning

    1. Subjects who are intending to father a child in the 90 days following the study or are unwilling to abstain from sexual intercourse with pregnant or lactating women.
    2. Subjects who are unwilling to use a condom/spermicide in addition to having their female partner use another form of contraception such as an IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or a tubal ligation if the woman could become pregnant from the time of the assessment visit until 3 months following the study.
11. Other; Non-removable metal objects such as metal plates, screws etc in their chest or abdominal area which in the opinion of the PMI or medically qualified designee/ responsible physician could affect the study conduct.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 9 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Site of release of radiolabel | To 14 hours post-dose
  Site of release of radiolabel determined by a qualified assessor based on gamma scintigraphy images
Time to release of radiolabel | To 14 hours post-dose
  Site of release of radiolabel determined by a qualified assessor based on gamma scintigraphy images
To visualise radiolabel dispersion within the colon | To 14 hours post-dose
  To visualise the disintegration and dispersion of delayed release tablets from gamma scintigraphy images of the colon

SECONDARY OUTCOMES:
Cmax | To 24 hours post-dose
  Maximum Plasma Concentration
Tmax | To 24 hours post-dose
  Time of Maximum Plasma Concentration
Tlag | To 24 hours post-dose
  Lag Time
AUClast | To 24 hours post-dose
  Area Under the Curve from time 0 to 24 hours
AUC0-inf | To 24 hours post-dose
  Area Under the Curve from time 0 to infinity
K | To 24 hours post-dose
  Terminal First Order Rate constant
t1/2 | To 24 hours post-dose
  Half Life
Adverse Events | 14 days
  Number of Participants With Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Howard Stevens, PhD, Principal Investigator — BDD Pharma Ltd
Locations (1):
- BDD Pharma Ltd, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No